CLINICAL TRIAL: NCT04868058
Title: Serratus Anterior Plane Block or Erector Spinae Plane Block Used as an Adjuvant for Hybrid Arrhythmia Ablation Surgery
Brief Title: Serratus Anterior or Erector Spinae Block for Hybrid Arrhythmia Ablation Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough patients were recruited
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: SAPB-ESPB hybrid AAS study
Record Dates: First submitted 2019-12-02; First posted 2021-04-30 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Arrhythmia
Keywords: Arrhythmia; Ablation; Pain
MeSH Terms: conditions — Arrhythmias, Cardiac; Pain | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: This clinical investigation is an interventional uni-center, prospective, open, randomized, double arm, blinded to the pain physician and the patient, clinical evaluation
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 1 AF SAPB (Experimental): Atrial fibrillation. Serratus anterior plane block
  Interventions: Drug: Ropivacaine injection
- 2 AF ESPB (Experimental): Atrial fibrillation. Erector spinae plane block
  Interventions: Drug: Ropivacaine injection
- 3 VT SAPB (Experimental): Ventricular Tachycardia.Serratus anterior plane block
  Interventions: Drug: Ropivacaine injection
- 4 VT ESPB (Experimental): Ventricular Tachycardia. Erector spinae plane block
  Interventions: Drug: Ropivacaine injection
- 5 ISNT SAPB (Experimental): Inappropriate Sinus node tachycardia. Serratus anterior plane block
  Interventions: Drug: Ropivacaine injection
- 6 ISNT ESPB (Experimental): Inappropriate Sinus node tachycardia. Erector spinae plane block
  Interventions: Drug: Ropivacaine injection

INTERVENTIONS:
Drug: Ropivacaine injection — Ropivacaine : 0.4 ml/kg (ideal body weight!) of 5mg/ml (20 to 30 ml bolus dose (100-150 mg), maximum dose 200 mg ropivacaine
  Other Names: Naropin

SUMMARY:
The purpose of this study is to evaluate differences between single-shot EQUAL ropivacaine doses of the serratus anterior plane block (SAPB) or erector spinae plane block (ESPB) injection, when used as adjuvant to treat postoperative pain, after one-stage unilateral hybrid arrhythmia (atrial fibrillation, ventricular tachycardia, inappropriate sinus node tachycardia) ablation surgery. The primary outcomes are to evaluate block placement efficacy in the hybrid surgery setting (total time to block placement in seconds, time to visualization of location of injection in seconds, adequacy of ropivacaine spread) by picturing and worst numerical scale pain at rest or moving, using a visual analog pain scale from 0= no pain to 10= maximal pain, in the first 12 hours after admission to the post-anaesthesia care unit. Secondary outcomes aim to evaluate to investigate pain location, additional analgesic consumption and requests, ease of breathing, breathing quality, sleeping quality and quantity, duration of hospitalisation, and general level of satisfaction.

DETAILED DESCRIPTION:
This clinical investigation is an interventional uni-center, prospective, open, randomized, double arm, blinded to the pain physician and the patient, clinical evaluation.

To ensure the same number of patients in each group, a stratified block randomization will be performed. A randomization list is generated for each type of arrhythmia. Patients will be block randomized into two groups: the serratus anterior plane block (SAPB) arm or the erector spinae plane block (ESPB) arm. As such the nerve block performing physician will be informed on the nerve block choice just before surgery.

132 consecutive patients. (22 in each group) Single Center study: Universitair Ziekenhuis Brussel - department of Anesthesiology 3 years Subject will be followed till 3 days post-procedure

Primary outcome measurement details:

The total time to block placement is obtained by starting a timer after local antiseptic application, just before puncturing the skin, to full injection of the local anaesthetic ropivacaine where the timer will be stopped.

In practice: a physician places the nerve block, a nurse anaesthetist manages the patient and a second nurse assistant records the timing and takes a picture just before drug injection and after block injection The time to visualization of the optimal location before nerve block injection is defined as the time needed to find the best place before local anaesthetic injection.

A picture of the location will be taken just before and after injection (by the second nurse assistant with an I-phone or similar device and kept with the patient's file Pain assessment will start 1 h after ICU admission by a different team (ICU nurse- intensive care physician or pain nurse). The first 24h assessments are blinded to the block performing physician.

Visual- analog- pain scores (0 no pain-10= maximal pain) will be analysed at rest or moving every 4 h or more depending on the patient's needs/requests for the first 24 h. After this period pain will be analysed twice daily (morning and afternoon) up to 72 h after start of surgery or less when dismissed earlier.

Secondary outcome measurements will be recorded after the initial 24h twice/da (morning and afternoon) by a pain nurse. Written data will be transmitted for storage to REDCAP.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years.
2. Provision of signed informed consent prior to any study-specific procedure
3. Selected for Hybrid Rhythm ablation surgery (ISNT, VT, AF)
4. American Society of Anesthesiologist physical Status I to III
5. Dutch, French or English speaking
6. Ability to follow the study protocol
7. BMI > 35 kg/m2 . BMI or Body mass index will be obtained from body weight in kg divided by the square of the length in meter and is expressed in kg/m2

   -

   Exclusion Criteria:
   * a. History of chronic pain or drug treatment abuse
   * b. Depression, psychiatric morbidity or mal-adaptive coping behaviour
   * c. Neuropathy
   * d. Severe anxiety or other mental ailment, taking drugs affecting their capacity to assess pain (gabapentin, pregabalin, opiod use)
   * e. Chronic or acute skin infection of the back or the lateral thorax
   * f. Hypersensitivity to ropivacaine
   * g. Severe hepatic, renal , pulmonary or cardiac (EF < 30%) disease or refuse to participate to the study..

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
evaluate block placement efficacy in the hybrid surgery setting specifically time to placement in seconds | Time to placement: 1200 seconds
  Time to placement in seconds
evaluate block placement efficacy in the hybrid surgery setting visualization time of location of injection by picturing | Visualisation is done by picturing to confirm adequate block (up 120 seconds)
  visualisation time of location of injection
evaluate block placement efficacy in the hybrid surgery setting adequacy of ropivacaine spread by picturing | picturing Confirms time of block placement (up to 300 seconds)
  Block placement efficacy by seeing the ropivacaine spread
Worst numerical scale pain in the first 12 h after admission to the post-anaesthesia care unit. | 12 hours
  Maximal pain assesed by visual analog scale ,where 0= no pain 10= maximal pain

SECONDARY OUTCOMES:
Pain location | 72 hours
  Place of pain: sternal; back, thorax, shoulder, throat, neck
Additional analgesic consumption and requests | 72 hours
  Pain drugs used: paracetamol in grams, piritramide in milligrams, diclofenac in milligrams, aspirin in milligrams, colchicine in grams
Ease of breathing, breathing quality | 72 hours
  Breathing evaluation: superficial, tense, normal, deep
Sleeping quantity | 72 hours
  Number of hours slept after surgery
Duration hospital Stay | From 2 to 15 days
  Length of hospital stay
Body Mass Index | Will be assessed on screening day or exported up to 2 weeks before screening day.
  BMI or Body mass index is obtained from body weight in kg divided by the square of the length in meter) and is expressed in kg/m2).Exclusion criteria if above > 35 kg/m2
Ideal body weight | Will be assessed on screening day or exported up to 2 weeks before screening day.
  Ideal body weight will be calculated from body weight in kg, length in cm and gender on https://by globalrph.com/medcalc. It is expressed in kg and used for drug dosing

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis, Brussels, Brussels Capital, Belgium